CLINICAL TRIAL: NCT06322524
Title: Shanxi Key Laboratory of Artificial Intelligence Assisted Diagnosis and Treatment for Mental Disorder
Brief Title: Study on Gamma Sensory Flicker for Insomnia
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Shanxi Medical University (Other)
Collaborators: Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Yong Xu, Clinical Professor, The First Affiliated Hospital of Shanxi Medical University
Other Study IDs: FirstShanxiMU_jsk
Record Dates: First submitted 2024-03-05; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Sleep Quality; Sleep Duration; Sleep Onset Latency
Keywords: gamma sensory flicke; insomnia; sleep quality; adherence; adverse effect
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- insomnia group: insomnia participants participants underwent polysomnography (PSG), the Insomnia Severity Index (ISI), the Pittsburgh Sleep Quality Index (PSQI), the Self-Rating Anxiety Scale (SAS), and the Self-Rating Depression Scale (SDS). prior to the commencement of the study.
  8 weeks of the intervention of Gamma sensory flicker, 30 min per day. After 8 weeks study, participants underwent polysomnography again. In the first week of study, participants were required to keep a daily sleep diary everyday.
  In the eighth week of study ,participants were required to keep a daily sleep diary everyday.
  Interventions: Device: Gamma sensory flicker

INTERVENTIONS:
Device: Gamma sensory flicker — participants were exposed to flicker stimulation through a light and sound device, the flicker was 40 Hz.

SUMMARY:
This prospective observational study enrolled adult volunteers for a sleep quality research study through a questionnaire survey distributed via a WeChat two-dimensional code from May 2021 to April 2022. Participants were exposed to flicker stimulation through a light and sound device for a duration of 8 weeks with daily monitoring.

DETAILED DESCRIPTION:
This prospective observational study enrolled adult volunteers for a sleep quality research study through a questionnaire survey distributed via a WeChat two-dimensional code from May 2021 to April 2022. Participants were exposed to flicker stimulation through a light and sound device for a duration of 8 weeks with daily monitoring.

A total of 37 participants underwent polysomnography (PSG) prior to the commencement of the study.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of insomnia according to DSM-5 Cumulative score of ≥7 on the seven-factor components of the Pittsburgh Sleep Quality Index. Sleep disturbances manifest at least three times per week.

Exclusion Criteria:

Secondary insomnia related to other mental disorders Substance-induced sleep disorders Environmental sleep disorders Sleep apnea syndrome. Stroke patients Insomnia caused by physical diseases, Severe ophthalmic diseases Brain tumors Suspected or confirmed history of alcohol or drug abuse Psychoactive drugs Pregnancy Previous participation in clinical trials within the past three months Epilepsy or family history of epilepsy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 to 70, of any gender, must have completed at least primary school education with a minimum of 5 years of schooling, possess the ability to comprehend instructional language, willingly provide informed consent, and demonstrate adherence to the research protocol.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Treatment adherence rate | 8 weeks （56 days）
  Participants adhered well to flicker therapy over eight weeks, as measured by the percentage of days they used the device out of the total days they were assigned to use it.
  Treatment adherence rate = days the patient completed treatment on time/56 days×100%
Patient treatment adherence rate | 8 weeks （56 days）
  Participants adhered well to flicker therapy over eight weeks, as measured by the percentage of days they used the device out of the total days they were assigned to use it.
  Patient treatment adherence rate = sum of all treatment adherence rates / number of patients participating in treatment×100%
Incidence rate of adverse reaction | 8 weeks
  Describe the specific situation of adverse reactions, including types, frequency, severity, and whether they have been relieved.
  Incidence rate of adverse reactions = number of people experiencing adverse reactions/total number of people participating in treatment x 100%
Differences in sleep duration between the first and eighth weeks | 8 weeks
  Keep sleep diaries for the first and eighth weeks of treatment.
  A comparison of average sleep duration （hour） between the first and eighth weeks of treatment.
Differences in sleep onset latencies between the first and eighth weeks | 8 weeks
  Keep sleep diaries for the first and eighth weeks of treatment.
  A comparison of average sleep onset latencies （min）between the first and eighth weeks of treatment.
Differences in awakening times between the first and eighth weeks | 8 weeks
  Keep sleep diaries for the first and eighth weeks of treatment.
  A comparison of average waking times （times） between the first and eighth weeks of treatment.

SECONDARY OUTCOMES:
pre-sleep efficiency. | pre-intervention
  Sleep efficiency=total sleep time/total bed rest time x 100% according to the Polysomnography.
post-sleep efficiency. | 8 weeks
  Sleep efficiency=total sleep time/total bed rest time x 100% according to the Polysomnography.

CONTACTS AND LOCATIONS:
Locations (1):
- Yong Xu, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
We will share individual participant data (including informed consent) after the study was published

REFERENCES:
- [Background] Son G, Neylan TC, Grinberg LT. Neuronal and glial vulnerability of the suprachiasmatic nucleus in tauopathies: evidence from human studies and animal models. Mol Neurodegener. 2024 Jan 10;19(1):4. doi: 10.1186/s13024-023-00695-4. PMID 38195580
- [Background] Fernandez-Ruiz A, Oliva A, Soula M, Rocha-Almeida F, Nagy GA, Martin-Vazquez G, Buzsaki G. Gamma rhythm communication between entorhinal cortex and dentate gyrus neuronal assemblies. Science. 2021 Apr 2;372(6537):eabf3119. doi: 10.1126/science.abf3119. PMID 33795429
- [Background] Martorell AJ, Paulson AL, Suk HJ, Abdurrob F, Drummond GT, Guan W, Young JZ, Kim DN, Kritskiy O, Barker SJ, Mangena V, Prince SM, Brown EN, Chung K, Boyden ES, Singer AC, Tsai LH. Multi-sensory Gamma Stimulation Ameliorates Alzheimer's-Associated Pathology and Improves Cognition. Cell. 2019 Apr 4;177(2):256-271.e22. doi: 10.1016/j.cell.2019.02.014. Epub 2019 Mar 14. PMID 30879788
- [Background] Manippa V, Palmisano A, Filardi M, Vilella D, Nitsche MA, Rivolta D, Logroscino G. An update on the use of gamma (multi)sensory stimulation for Alzheimer's disease treatment. Front Aging Neurosci. 2022 Dec 15;14:1095081. doi: 10.3389/fnagi.2022.1095081. eCollection 2022. PMID 36589536
- [Result] Lucey BP. It's complicated: The relationship between sleep and Alzheimer's disease in humans. Neurobiol Dis. 2020 Oct;144:105031. doi: 10.1016/j.nbd.2020.105031. Epub 2020 Jul 29. PMID 32738506